CLINICAL TRIAL: NCT05055791
Title: A Phase Ⅰ/Ⅱ Study to Evaluate the Safety, Tolerance, Pharmacokinetics and Efficacy of SYHX1903 in Patients With Relapsed/Refractory Hematologic Malignancies
Brief Title: A Study to Evaluate the Safety and Tolerance of SYHX1903 in Patients With Relapsed/Refractory Hematologic Malignancies
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYHX1903-CSP-001
Record Dates: First submitted 2021-08-11; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-08

CONDITIONS: Acute Myeloid Leukemia; Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Lymphoma; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Cohort 1-3 dose level 1-3 in subjects with relapsed or refractory haematological malignancies including AML/ALL/CMML/CLL.
  Interventions: Drug: SYHX1903
- Arm 2 (Experimental): Cohort 1-3 dose level 1-3 in subjects with relapsed or refractory haematological malignancies including AML/ALL/CMML/CLL.
  Interventions: Drug: SYHX1903

INTERVENTIONS:
Drug: SYHX1903 — SYHX1903 tablets, orally, qd

SUMMARY:
This trial is an open-label, multi-center, dose escalation, dose expansion, and cohort expansion phase I/II clinical study of SYHX1903 in patients with relapsed/refractory hematologic malignancies. This trial aims to evaluate the safety, tolerance, pharmacokinetics, and preliminary antitumor activity of SYHX1903 in patients with relapsed/refractory hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed/refractory hematologic malignancies confirmed by the World Health Organization (WHO) criteria.
* Eastern Cooperative Oncology Group (ECOG) score ≤ 1.
* Life expectancy ≥ 3 months.

Exclusion Criteria:

* Pregnant and lactating females.
* Proven hematologic malignancies of the central nervous system.
* Diagnosed acute promyelocytic leukemia (predominantly granulocytic promyelocytes in bone marrow, which are ≥ 30% in NEC).
* History of other malignant tumors within 5 years, except for cured skin basal cell carcinoma, skin squamous cell carcinoma or cervical carcinoma in situ.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2021-12-29 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities | 28 days
  DLTs will be determined from monitoring adverse events (AEs), and abnormal laboratory tests (clinical chemistry, hematology, and urinalysis), physical examinations, vital signs (blood pressure and pulse), and electrocardiogram (ECG).
Incidence of adverse events | 1 year
  Number of subjects with adverse events as a measure of safety and tolerability including changes in vital signs, electrocardiograms (ECGs), safety and laboratory parameters
Antitumor activity of SYHX1903 in patients by assessing overall response rate (ORR) | 1 year
  To assess proportion of patients with anti tumor response to SYHX1903. response assessment by Cheson (2014) criteria and myeloma (Palumbo 2014) Response will be evaluated every 4-12 weeks (based on disease type) until progression

IPD SHARING:
Plan to Share IPD: No